CLINICAL TRIAL: NCT02024139
Title: Efficacy of Chewing Sugarless Gum for Reduction of Orthodontic Fixed Appliance Activation Pain
Brief Title: Efficacy of Chewing Sugarless Gum for Reduction of Orthodontic Appliance Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Athbi Alqareer, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DD01/13
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Pain Associated With Fixed Orthodontic Treatment
Keywords: Orthodontic pain; Chewing gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chewing Sugarless Gum and Mouthwash (Experimental): Patients are asked to chew sugarless gum 3 times per day in addition to using a fluoridated mouthwash 3 times per day
  Interventions: Other: Chewing Sugarless Gum; Other: Using Mouthwash
- Using fluoridated mouthwash (Placebo Comparator): Using Mouthwash: Patients are asked to use a fluoridated mouthwash 3 times per day as a placebo
  Interventions: Other: Using Mouthwash

INTERVENTIONS:
Other: Chewing Sugarless Gum — Chewing sugar free gum three times per day for 5-10 minutes
  Other Names: Mentos 3D sugar free gum
  Arms: Chewing Sugarless Gum and Mouthwash
Other: Using Mouthwash — Rinse mouth with plax sensitive fluoridated mouthwash for 30 seconds, three times per day
  Other Names: Place fluoridated mouthwash

SUMMARY:
This study investigates whether chewing sugar-free chewing gum can reduce pain associated with braces treatment. The study collects pain scale records for 10 consecutive days after placement of braces. No changes to patients routine braces treatment is done. All materials used are available over the counter.

DETAILED DESCRIPTION:
Objectives:

1. To characterize the intensity and dynamics of pain experienced by patients following orthodontic appliance placement and activation using a set of Visual Analogue pain scale diaries
2. To determine whether chewing sugarless gum 3 times per day (and using a non-analgesic mouthwash) reduces orthodontic pain compared to only using a mouthwash (placebo)

Importance:

Pain from orthodontic treatment affects most if not all orthodontic patients. Learning more about the nature and timing of pain will help clinicians give patients a more scientific, evidence-based informed consent. If chewing gum was found to reduce pain, then we would have validated a common clinical advice with scientific evidence. We will also have established a non-pharmacological option for pain reduction with orthodontic treatment. If chewing gum was not found to reduce pain (or was found to increase it), then we can advise our patients against using it and advise clinicians against recommending it.

Research Methodology

Inclusion criteria:

* Comprehensive fixed upper and lower orthodontic treatment scheduled
* Age of patient between 10-35

Exclusion Criteria:

* Partial engagement of teeth
* The use of functional or extra-oral appliances
* Patients on regular pain medications
* Patient experiencing chronic pain
* Patients unable to consume sugarless gum because of health reasons e.g. phenyl ketone urea o Patients with mental or cognitive impairments

Group Assignment:

For our sample size estimation we used a standard deviation of 20 (taking into consideration several previous studies of other investigators), an effect size of 15, a significance level of 0.05, and a power of 0.8. It indicates the need for 58 subjects in total. Based on this, our goal is to include 80 subjects in anticipation of possible drop-outs. Patients will be randomly assigned to one of two groups: a chewing gum group and a control mouthwash group. Study kits will be numbered according to a random number table. Forty kits will contain instructions and supplies for the chewing gum group and forty will contain instructions and supplies for the control group. Assignment is done immediately after orthodontic appliances are placed. Operators will be blinded to the group assignment as it is done by a separate investigator. This investigator will administer to the patients the consent forms and give them instructions according to their group assignment. The investigator will give the participants a pre- randomized study kit containing a VAS booklet and either enough servings of chewing gum and a container of mouthwash or a container of mouthwash only with corresponding verbal and written instructions.

Materials used:

We will provide to the chewing gum group subjects with enough servings of Wrigley's extra sugar-free chewing gum (with some extra pieces as backup). The chewing gum used is Mentos 3D which contains both sorbitol and xylitol (non-hard coated type used). The mouth wash used for both groups is Plax SensitiveTM fluoride containing mouthwash which is alcohol free and causes significantly less burning sensations than regular mint mouthwashes. The mouthwash will be supplied to the subjects in unlabeled containers so as to work as a placebo. The subjects will not be told that this is a regular mouthwash with no pain reducing effects. Each of the two groups' subjects are ignorant to what the other group is receiving and whether they are in a control group or not.

The VAS pain scale:

The VAS pain scale used in the study comprises a 100mm horizontal line where one end indicates "no pain" and the other end indicates "worst possible pain". The patients will mark each pain scale after fitting their teeth together. During the first day, patients will mark a scale every 3 hours until bedtime starting immediately after appliance placement. For the following 9 days, patients will mark 2 pain scales per day, one scale when they wake up and one at bedtime. The patient places a mark on the scale according to their judgment of the amount of pain they experience. The response is then measured to the nearest 0.5mm and can be used as pseudo-numerical data.

The VAS booklet:

Booklets are uniquely identified by a serial number and the patients phone number. Each booklet will be pre-randomized and assignment to either the gum group or the control group. The group assignment and serial number are indicated on the booklet cover. After instructions are given, the booklet cover is removed and kept in a closed container. The group assignment is only initially known to the investigator who administers the instructions. The remaining pages of the booklet will only be identified by the serial number of the participant with no mention of the group assignment. This way the group assignment is kept secret from both the operators who place the appliances, and the measurement investigator who will later measure the patients' responses. The booklet will contain space for participants to indicate if they have taken any non-study related medication (e.g. an analgesic). A copy of the booklet is included will this document.

Blinding:

The design of the study is double blinded. Operators placing the appliances do not know which group the patient belongs to because assignment is done after appliance placement. The investigator measuring the patient responses does not know the group assignment because it is not indicated on the VAS booklet. The patients can be considered to be blinded because they are not aware of what the other group is receiving or that they are using a standard mouthwash that does not affect pain. After all measurement are done the booklet covers are reunited with their respective booklets for statistical data analysis.

Patient Compensation:

Patients will receive an electric toothbrush as an incentive for completing the study.

ELIGIBILITY:
Inclusion Criteria:

* fixed upper and lower orthodontic appliance therapy scheduled

Exclusion Criteria:

* tooth extractions within one week
* chronic pain
* regular use of analgesics
* partial appliance engagement
* use of extra-oral appliances like headgear
* patients unable to consume sugarless gum like phenylketonuria patients

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain scale reading | 10 days
  Patients mark a 100mm visual analog pain scale to rate tooth pain experienced during the first 10 days of their routine orthodontic treatment

SECONDARY OUTCOMES:
Patient subjective assessment of pain experience | 10 days
  Patients answer subjective questions about pain experience and whether is affects their decision to undergo orthodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Athbi Alqareer, BDM, DMSc, Principal Investigator — Kuwait University
Locations (1):
- Bneid Algar Dental Speciality Center, Kuwait City, Kuwait, Kuwait